CLINICAL TRIAL: NCT06497894
Title: No More Sleepless Nights in Perimenopause - an Open Label, Randomized, Parallel-group, Active Controlled Intervention Study in Perimenopausal Women With Vasomotor Symptoms and Insomnia to Investigate the Efficacy of Hormone Replacement Therapy and Cognitive Behavioral Therapy
Brief Title: No More Sleepless Nights in Perimenopause
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00209
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Insomnia; Menopause
Keywords: Perimenopause; Insomnia; Cognitive Behavioral Therapy; Hormone Replacement Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Hormone Replacement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioral Therapy for insomnia (CBT-I) (Experimental): Participants in this experimental arm will receive cognitive behavioral therapy specifically designed to treat insomnia (CBT-I). The therapy will be delivered over 8 weekly sessions, each lasting 60 minutes. The sessions will include techniques such as sleep restriction, stimulus control, cognitive restructuring, and relaxation training. The primary goal is to improve sleep quality and reduce the severity of insomnia.
  Interventions: Behavioral: Cognitive Behavioural Therapy for Insomnia (CBT-I)
- Hormone Replacement Therapy (HRT) (Active Comparator): Participants in this experimental arm will receive hormone replacement therapy, specifically a combination of estrogen and progesterone over the course of 8 weeks. The therapy aims to alleviate menopausal symptoms, including insomnia, by addressing hormonal imbalances.
  Interventions: Drug: Hormone Replacement Therapy (HRT)
- Sleep Hygiene (Sham Comparator): Participants in this sham comparator arm will receive sleep hygiene instructions. Instructions will be delivered over 8 weekly sessions. The instructions will provide general information about healthy sleep habits, such as food and drink choices, a regular sleep schedule, evening routine, etc. Although being widely used in daily clinical practice, sleep hygiene shows no significant effect as monotherapy in patients with an established insomnia. The sleep hygiene condition in this study is matched to CBT-I in frequency and intensity of contact.
  Interventions: Behavioral: Sleep Hygiene

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Insomnia (CBT-I) — CBT-I is conducted in an individual setting according to the manual used in McCurry (1). Factors at the level of behavior, cognitions, and physiology that perpetuate sleep onset and sleep maintenance disorders are addressed. In addition, psychoeducation on sleep and sleep hygiene, stimulus control, sleep restriction, relaxation, structured worry time, cognitive restructuring, and relapse prevention are part of the training. Each session will include homework.
  Arms: Cognitive Behavioral Therapy for insomnia (CBT-I)
Drug: Hormone Replacement Therapy (HRT) — Standard-dose continuously-combined bio-identical HRT containing transdermal estradiol 1.5 mg/d (= 2 strokes of Oestrogel® Dispenser) and oral micronized progesterone (= 1 capsule of Utrogestan® 200). This combination is the most popular HRT regimen, as it has a neutral effect on lipids, glucose, haemostasis. Participants will receive a conventional prescription for the 2 products that are covered by all health insurances in Switzerland.
  Arms: Hormone Replacement Therapy (HRT)
Behavioral: Sleep Hygiene — Sleep hygiene refers to healthy sleep habits, e.g. food and drink choices, a regular sleep schedule, evening routine. Although being widely used in daily practice, sleep hygiene shows no significant effect as monotherapy in patients with an established insomnia. The sleep hygiene condition in this study is matched to CBT-I in frequency and intensity of contact.
  Arms: Sleep Hygiene

SUMMARY:
The goal of the clinical trial is to learn if Hormone Replacement Therapy (HRT) and Cognitive Behavioral Therapy (CBT-I) can treat insomnia in menopausal women. The main questions it aims to answer are:

* Are HRT and CBT-I effective in reducing insomnia in menopausal women?
* Are HRT and CBT-I comparable in terms of reducing insomnia severity in this population?

Researchers will compare HRT and CBT-I to an active control group, receiving sleep hygiene instructions.

Participants will:

* Complete a screening and baseline assessment
* Receive Hormone Replacement Therapy (as prescribed), Cognitive Behavioral Therapy (1/week), or sleep hygiene instructions (1/week) for 8 weeks.
* Keep a daily diary (sleep e-diary), to assess sleep-quality.
* Wear an electroencephalogram (EEG) during 6 nights (3 at baseline & 3 post-intervention), to assess deep sleep cycles and waking episodes.
* Receive a phone call for intervention compliance
* Complete a post-intervention assessment.

ELIGIBILITY:
Inclusion Criteria:

* Late menopausal transition according to Stages of Reproductive Aging criteria (STRAW+10)
* Pittsburgh Sleep Quality Index (PSQI) score > 5
* Insomnia Severity Index (ISI) score > 7
* Somato-vegetative domain of the Menopause Rating Scale (MRS)-II ≥ 4 points
* Willingness to use HRT for menopausal symptom reliefs

Exclusion Criteria:

* Other sleep-wake disorders according to DSM-5, assessed with validated questionnaires (Sleep-Health Questionnaire, Epworth Sleepiness Scale (ESS))
* Untreated hormonal disorder
* Obesity (BMI ≥ 30)
* Current psychotherapy
* Current psychopharmacological therapy including regular sleep medication
* History of unsuccessful CBT-I
* Psychiatric illness
* Substance abuse (≥ 7 cigarettes/day, no more than 2 standard WHO drinks per day, other drugs)
* Shift work
* Long-haul flights across different time zones in the past 3 months
* Pregnancy and lactation
* Contraindications to HRT according to drug information (https://www.swissmedicinfo.ch/)
* Inability to follow procedures or insufficient knowledge of project language
* Inability to give consent

Ages: 45 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of Insomnia Severity | Week 10
  Change from baseline in Insomnia Severity Index (ISI). The ISI is a seven-item questionnaire, asking respondents to rate the severity of sleep-related symptoms on 5-point Likert scales (Ranging between 0 = not applicable and 4 = very strong). Total values may range between 0 and 28, where 0 indicates no presence of sleep-related symptoms and 28 indicates very severe symptoms.

SECONDARY OUTCOMES:
Improvement in Climacteric Syndrome | Week 10
  Change from baseline in Menopause Rating Scale (MRS-II) The MRS-II is an eleven-item questionnaire, asking respondents to rate the severity of climcteric syndrome-related symptoms on 5-point Likert scales (Ranging between 0 = not applicable and 4 = very strong). Total values may range between 0 and 44, where 0 indicates no presence of symptoms and 44 indicates very severe symptoms.
Changes in bio-functional age | Week 10
  Change from baseline in biofunctional status (i.e. differences between chronological age and biofunctional age).
Changes in maladaptive sleep-related cognitions | Week 10
  Change from baseline in Dysfunctional Attitudes and Beliefs about Sleep Scale (DBAS).
  The DBAS is a sixteen-item questionnaire, asking respondents to rate their attitudes/beliefs about sleep on 10-point numerical rating-scales (discrete intervals), ranging between 0 (I do not agree at all) and 10 (I agree completely). Total values may range between 0 and 160, where 0 indicates no presence of dysfunctional attitudes and 160 indicates very severe levels of maladaptive sleep-related cognitions.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Stute, Prof., Principal Investigator — University Hospital of Bern, Department of Gynecological Endocrinology & Reproductive Medicine
Locations (1):
- University Hospital of Bern, Department of Gynecological Endocrinology & Reproductive Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavicic E, Stute P, Rudzik F, Urech A, Lozza-Fiacco S. No more sleepless nights in perimenopause-an open-label, randomized, parallel-group, active controlled intervention study in perimenopausal women with vasomotor symptoms and insomnia to investigate the efficacy of hormone replacement therapy and cognitive behavioral therapy for the treatment of insomnia: study protocol. Trials. 2025 Dec 30. doi: 10.1186/s13063-025-09366-9. Online ahead of print. PMID 41462320